CLINICAL TRIAL: NCT06080087
Title: Implementation Toolkit to Enhance EBP Among Marginalized Families
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, James Lee, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004246
Record Dates: First submitted 2023-07-09; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Autism; Early Intervention
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be blinded into which condition they were assigned into
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group will receive access to the I-TEAM
  Interventions: Behavioral: I-TEAM
- Waitlist control (No Intervention): Waitlist control group will not receive access to the I-TEAM until the Intervention group has completed the 8-week intervention.

INTERVENTIONS:
Behavioral: I-TEAM — I-TEAM is a web-based implementation toolkit that supports to enhance cultural responsiveness of EI providers in their EBP delivery with minoritized families of young autistic children
  Arms: Intervention

SUMMARY:
Although the efficacy of early intervention (EI) for autistic children and their families has been established, many marginalized families with diverse cultural and linguistic backgrounds still report inequitable access to evidence-based practices (EBP). There are several strategies to increase EBP implementation that are especially relevant to marginalized families who report inequitable access to coaching from EI providers, such as increasing the capacity of EI providers to coach families in a culturally responsive way. However, EI providers are provided with limited professional development in both family coaching and cultural responsiveness, which results in perpetuation of EBP implementation failure. Thus, it is crucial to develop and validate an implementation toolkit that comprises strategies to enhance cultural responsiveness in the uptake of EBPs among EI providers. Therefore, the overall purpose of this research is to identify facilitators and barriers of EBP implementation among marginalized families in EI to aid the development an implementation toolkit with a focus on capacity building of EI providers to implement EBP with cultural responsiveness. This will involve conducting individual interviews with EI providers.

ELIGIBILITY:
There are two sets of inclusion criteria for both types of participants.

Inclusion Criteria for EI providers:

* Currently working with minoritized families of young children within Part-C
* Willing to complete I-TEAM as instructed
* Over the age of 18

Exclusion Criteria for EI providers:

* Not able to complete I-TEAM as instructed

Inclusion Criteria for families:

* Having a minoritized backgrounds (e.g., migrant/refugee background, primarily speaks another language other than English at home)
* Having a young child eligible for early intervention services

Exclusion Criteria for EI providers:

* Not currently receiving early intervention services

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Coaching Fidelity Scale (CFS) | Change from baseline at 8 weeks
  CFS is an observational measure to assess coaching fidelity during an interaction between a coach and a learner
Cultural Self-Efficacy Scale for Early Interventionists (CSES-EI) | Change from baseline at 8 weeks
  CSES-EI is a 32-item, self-reported measure of cultural self-efficacy of early intervention providers
Social Validity | Change from baseline at 8 weeks
  We will measure acceptability and feasibility of I-TEAM

SECONDARY OUTCOMES:
Measure of NDBI Strategy Implementation: Caregiver Change (MONSI-CC) | Change from baseline at 8 weeks
  MONSI-CC is an observational measure that detects changes in caregivers' use of NDBI strategies in early intervention
Autism-specific parenting self-efficacy | Change from baseline at 8 weeks
  We will use this self-reported tool to assess self-efficacy of parents of young autistic children
Social validity | Change from baseline at 8 weeks
  We will assess social validity, including satisfaction with their services, reports of cultural responsiveness of their providers, acceptability of early intervention among intervention recipients

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No